CLINICAL TRIAL: NCT05110664
Title: A Double-blind, Cross-over, Placebo-controlled, Proof-of-concept Study Using Oral Peptide YY3-36 Solution to Investigate the Mechanistic Role of Lingual PYY in Regulating Appetite, Energy Intake and Food Preference in People With Overweight/Obesity
Brief Title: APPETITE: linguAl PYY3-36 on aPpEtite and acuTe Energy InTakE
Acronym: APPETITE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Collaborators: Gila Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 142589
Record Dates: First submitted 2021-09-24; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: obesity; appetite
MeSH Terms: conditions — Obesity | interventions — peptide YY (3-36)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort/Intervention 1: Meal test
  Interventions: Drug: PYY (3-36) Peptide; Drug: Placibo
- Cohort/Intervention 2: Ad libitum meal
  Interventions: Drug: PYY (3-36) Peptide; Drug: Placibo

INTERVENTIONS:
Drug: PYY (3-36) Peptide — oral PYY3-36 solution
Drug: Placibo — oral placebo solution

SUMMARY:
A double-blind, cross-over, placebo-controlled, proof-of-concept study using oral peptide YY3-36 solution to investigate the mechanistic role of lingual PYY in regulating appetite, energy intake and food preference in people with overweight/obesity. The aim of this study is to investigate the mechanistic role of lingual PYY in regulating appetite, energy intake and food preference in people with overweight/obesity.

DETAILED DESCRIPTION:
In order to address the study objective two independent investigations in two separate groups of participants will need to be undertaken, to avoid cross-contamination of the results.

1. Cohort/Investigation 1: A randomised within-subject double-blind cross-over placebo-controlled study to investigate the role of lingual PYY in regulating fasted and post-meal appetite following a fixed energy intake meal.
2. Cohort/Investigation 2: A randomised within-subject double-blind cross-over placebo-controlled study to investigate the role of lingual PYY in regulating ad libitum energy intake and food preference.

People with overweight or obesity (BMI 25.0-39.9 kg/m2), identified via the University College London Hospitals (UCLH) Bariatric Centre for Weight Management and Metabolic Surgery and through advertising via University College London (UCL) and ULCH, will be invited to take part.

Potential participants will initially attend a screening visit, where informed, written consent will first be taken. During the screening visit, medical, drug and dietary histories will be taken and participant eligibility will be confirmed.

Participants will attend on two separate occasions at least 7 days apart for both cohort/investigation 1 and cohort/investigation 2. 20 participants per cohort/investigation will be randomised (in a 1:1 manner), stratified by sex, to receive either oral PYY3-36 solution or matched placebo at their first study visit. Participants will be recruited onto study/investigation 1 first and once this is complete, new subjects will be enrolled onto study/investigation 2.

Cohort/Intervention 1: The day prior to each visit participants will complete a 24 hour food diary and appetite scores at home. Participants will fast overnight (12 hours) and consume only water until reaching the clinical facility the following morning. Participants will need to refrain from exercise for 2 days prior to the study visits and from drinking alcohol. On arrival, medical history will be re-reviewed, sociodemographic information collected and a pregnancy test for women of childbearing potential will be performed. Body weight and composition will be measured. Baseline assessments of fasted subjective appetite assessed using validated visual analogue scales (VAS), saliva PYY levels (via saliva sample) and circulating gut hormones (via blood sample) will be taken.

A single dose of lingual PYY (GT-001) or placebo will be administered. Appetite scores and a paired blood and saliva sample will be collected 10-15 minutes later. 30 minutes after study drug application, participants will then be asked to consume a standardised fixed meal over 15 minutes using established protocol and appetite scores (VAS) and saliva and blood samples will be taken for 180 minutes post-meal at regular intervals. Participants will be asked to complete 24-hour food diary and appetite scores 6, 12 and 24 hours after the study visit.

Cohort/Intervention 2: The day prior to each study visit participants will complete a 24-hour food diary and appetite scores at home. Participants will fast overnight (12 hours) and consume only water until reaching the clinical facility the following morning. Participants will need to refrain from exercise for 2 days prior to the study visits and from drinking alcohol. On arrival, medical history will be re-reviewed, sociodemographic information collected and a pregnancy test for women of childbearing potential will be performed. Body weight and composition will be measured. Baseline assessments of fasted subjective appetite assessed using validated VAS, saliva PYY levels (via saliva sample) and circulating gut hormones (via blood sample) will be taken.

A single dose of lingual PYY (GT-001) or placebo will be administered. Appetite scores and a paired blood and saliva sample will be collected 10-15 minutes later. 30 minutes after study drug application, participants will be offered an extensive free-choice buffet lunch and asked to eat until full. Ad libitum energy intake and food preferences will be assessed. Participants will be asked to rank likeness of the items of the buffet. Appetite scores (VAS) and paired blood and saliva sample will be taken again 60 minutes from the onset of the meal. Participants will be asked to complete 24-hour food diary and appetite scores 24 hours after the study visit.

After a 7-day washout period participants in each cohort/intervention will be crossed-over and the same visit will be repeated. Both the participants and researchers will be blinded to the study condition.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults aged 18-65 inclusive. 2. People with a body mass index (BMI) between 25.0 and 39.9 kg/m2 3. Stable weight for past 3 months (≤5% change in preceding 3 months as reported by participants).

  4. Females of childbearing potential must be on highly effective contraception and have a negative pregnancy test within 7 days of their study visits. NOTE: Subjects are considered not of childbearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

  5. Fluent in English and able to understand and complete questionnaires. 6. Willing and able to provide written informed consent and comply with the study protocol.

Exclusion Criteria:

1. Female subjects who are pregnant or breast-feeding.
2. Female subjects of childbearing potential who are not on highly effective contraception.
3. Post-menopausal women who have not had a period of spontaneous amenorrhea for more than 1 year.
4. Previous bariatric surgery.
5. Type 1 or 2 diabetes.
6. Current use of weight loss medications or taking medication that affects appetite, e.g., antidepressants such as mirtazapine.
7. Food intolerances, or allergies, that would make fixed energy meal and/or ad libitum meal unable to be performed.
8. Impairment of sense of taste and/or smell, as per subject assessment and direct questioning.
9. Poor dental hygiene or oral pathology.
10. Current smokers of tobacco products.
11. Any other factor making the participant unsuitable in the view of investigator.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with overweight or obesity (BMI 25.0-39.9 kg/m2), identified via the University College London Hospitals (UCLH) Bariatric Centre for Weight Management and Metabolic Surgery and through advertising via University College London (UCL) and ULCH, will be invited to take part.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
appetite scores | up to 6 hours
  area-under-the curve for appetite scores. Not indicative of either bad or worse outcome, just subjective indication.
energy intake expressed as Kcal of eaten food | up to 6 hours
  ad libitum energy intake

SECONDARY OUTCOMES:
PYY levels | up to 6 hours
  Area-under-the-curve for saliva PYY levels
gut hormones levels | up to 6 hours
  Area-under-the-curve for gut hormones levels
24-h energy intake | 24 hours after study visit
24h appetite | 24 hours after study visit
  Subjective appetite scores for 24 hours following a fixed meal using VAS - a 1 to 10 scale will be used where the higher the score the higher the level of feeling of the item for the subject. No better or worse meaning applied a priory.
macronutrient selection | up to 1 hour
  Macronutrient content of consumed food during ad libitum meal
food preference using labelled magnitude scales (LMS) | through study completion, an average of 6 hours
  labelled magnitude scales (LMS) for components of the ad libitum meal
food preference questionnaire (FPQ) | once, at beginning of study visit
  The food preference questionnaire requires participants to rate their liking of 62 individual foods on a 5-point Likert scale, ranging from "not at all" to "a lot". A higher score indicative of greater liking of a food.